CLINICAL TRIAL: NCT01167075
Title: A Randomized, Prospective, Controlled, Double-blind, Single-center Pilot Study in Critically Ill Patients Investigating Tolerability and Efficacy of Low-volume Pharmaconutrition (Intestamin)
Brief Title: A Study in Critically Ill Patients Investigating Tolerability and Efficacy of Low-volume Pharmaconutrition (Intestamin)
Acronym: Intestamin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Schneider, Andrea MD, Medical School Hannover
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3941
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2005-12

CONDITIONS: Critical Illness; Adult; Sepsis; Systemic Inflammatory Response Syndrome
Keywords: critically ill; sepsis; antioxidants; enteral nutrition; SIRS (APACHE score 10-30); enteral feeding within 48 h of admission
MeSH Terms: conditions — Critical Illness; Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fresubin Original (Active Comparator)
  Interventions: Dietary Supplement: Fresubin Original
- Intestamin plus Fresubin Original (Experimental)
  Interventions: Dietary Supplement: Intestamin plus Fresubin Original

INTERVENTIONS:
Dietary Supplement: Fresubin Original
  Arms: Fresubin Original
Dietary Supplement: Intestamin plus Fresubin Original
  Arms: Intestamin plus Fresubin Original

SUMMARY:
The aim of the study is to assess the efficacy and tolerability of the low-volume supplement. The investigators randomized critically ill patients to receive Intestamin plus Fresubin or Fresubin alone.

DETAILED DESCRIPTION:
To compare early supplementation with antioxidants and glutamine using an enteral pharmaconutrition supplement (Intestamin®) to an energy adjusted standard elementary diet and to investigate its affect on clinical efficacy and tolerability in critically ill patients with sepsis/SIRS.

Methods: This was a prospective controlled randomized study in 58 critically ill patients. They received either Intestamin or a diluted Fresubin solution. After 10 or 14 days inflammatory parameters, catecholamine need, and maximal enteral delivery were determined.

ELIGIBILITY:
Inclusion Criteria:

* sepsis or SIRS (APACHE score 10-30),
* no severe gastrointestinal tract or metabolic diseases,
* enteral feeding within 48 h of admission,
* age 18-75 years,
* written consent by patient or next of kin. -

Exclusion Criteria:

* participation in a drug trial within the last 4 weeks before inclusion in this study,
* previous participation in this study,
* expected patient survival of less than 6 days,
* pregnancy or lactation,
* patients with unstable vital signs that would probably cause incidents that would make participation impossible or would lead to discontinuation,
* severe liver disease with cytolysis (ASAT >10 N) or impaired detoxification (ammonia >50 mmol/L, bilirubin > 50 μmol/L),
* gastrointestinal surgery in the last 4 weeks,
* severe enteritis/colitis,
* short intestine syndrome,
* gastrointestinal bleeding that requires intervention,
* patients who could not be enterally fed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Length of stay in ICU | 14 days
  The primary endpoints were length of stay in ICU and sufficient enteral feed.

SECONDARY OUTCOMES:
mortality | 14 days
  Secondary endpoints were APACHE score, days of fever, artificial ventilation, and antibiotics, mortality, catecholamine need, inflammation parameters (CRP, leukocytes, etc.), pneumonia with detection of bacteria, need for insulin, and length of hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School Hannover, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Schneider A, Markowski A, Momma M, Seipt C, Luettig B, Hadem J, Wilhelmi M, Manns MP, Wedemeyer J. Tolerability and efficacy of a low-volume enteral supplement containing key nutrients in the critically ill. Clin Nutr. 2011 Oct;30(5):599-603. doi: 10.1016/j.clnu.2011.04.003. Epub 2011 May 31. PMID 21621886